CLINICAL TRIAL: NCT03897517
Title: Effect of Proprietary Botanical Blend on Glycemic Control and Post-prandial Carbohydrate Absorption in Overweight, Insulin Resistant Adult Men and Women
Brief Title: Effect of Proprietary Botanical Blend on Glycemic Control and Post-prandial Carbohydrate Absorption
Acronym: PBPPCG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Plexus Worldwide (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 1355505-1
Record Dates: First submitted 2019-03-25; First posted 2019-04-01 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Hyperglycemia; Carbohydrate; Insulin Resistance; Malabsorption
Keywords: Glycemia; Carbohydrate blocker
MeSH Terms: conditions — Hyperglycemia; Insulin Resistance; Malabsorption Syndromes

STUDY DESIGN:
Intervention Model Description: Participants will receive both treatments in random order with a washout period of at least 1 week between the 2 study visits. Women will be measured during the follicular phase of the menstrual cycle.
Who Masked: Participant, Investigator
Masking Description: Treatment and placebo will be matched closely in color and appearance administered in a double blinded fashion as provided by the material supplier.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Proprietary Botanical Blend (Experimental): Proprietary Botanical Blend - Dietary supplement with alpha amylase and sucrase inhibitory activity. 2 capsules
  Interventions: Dietary Supplement: Proprietary Botanical Blend
- Placebo (Placebo Comparator): Non/minimally nutritive nonactive material: rice flour. 2 capsules
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Proprietary Botanical Blend — Oral administration of capsules containing proprietary botanical blend 30 minutes prior to carbohydrate ingestion.
  Arms: Proprietary Botanical Blend
Dietary Supplement: Placebo — Oral administration of capsules containing rice flour (placebo) 30 minutes prior to carbohydrate ingestion.
  Arms: Placebo

SUMMARY:
This project will test a unique botanical formula designed to inhibit alpha amylase (the primary starch degrading digestive enzyme) and inhibit sucrase (the primary sucrose degrading digestive enzyme) in order to reduce acute post prandial glycemia regardless of nutritive carbohydrate source.

DETAILED DESCRIPTION:
Type 2 diabetes is a metabolic disorder characterized by elevated fasting blood glucose and impaired insulin signaling (insulin resistance) and is associated with several comorbidities including neuropathy, retinopathy, kidney disease, and elevated risk for heart attack and stroke. Lifestyle interventions targeted towards prevention of type 2 diabetes include: maintaining and achieving healthy bodyweight, physical activity, avoiding tobacco use, and reducing sugar and saturated fat intake. The International Scientific Consensus Summit from the International Carbohydrate Quality Consortium indicated that diets low in glycemic index and glycemic load were important in the prevention and management of diabetes. Health supplements that can lower the glycemic index and glycemic load of food have potential to support the prevention of diabetes and improve blood glucose management by reducing post prandial glycemia and insulinemia. This project will test a unique botanical formula designed to inhibit alpha amylase (the primary starch degrading digestive enzyme) and inhibit sucrase (the primary sucrose degrading digestive enzyme) in order to reduce acute post prandial glycemia regardless of nutritive carbohydrate source. This proposal will fill a void in the literature by testing for the first time the effect of a combination of mulberry leaf, white kidney bean extract and cinnamon on postprandial carbohydrate absorption and glucose control in overweight, insulin resistant men and women. This project will provide pilot data to support larger studies, and studies to investigate long-term effects.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-65 years
* Men and women
* Able to provide written consent in English
* A body mass index between 23.0 and 30.0 kg/m2
* A fasting serum blood glucose level between 100.0 and 126.0 mg/dL

Exclusion Criteria:

* Current smoker
* Having a BMI less than 23.0 kg/m2 and higher than 30.0 kg/m2
* Having a fasting blood glucose level less than 100.0 mg/dL and higher than 126.0 mg/dL
* Suffering from known serious cardiac, hepatic, renal, pulmonary, gastrointestinal, endocrine or hematological disease based on investigator determination, aside from pre-diabetes
* Currently pregnant or breastfeeding
* Consuming more than 2 alcoholic drinks per day on average.
* Weight loss of more than 5% of body weight over the past 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-08-30 (Estimated); Primary Completion 2019-11-30 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Post Prandial Glycemia | 3 weeks
  Plasma glucose concentrations after the ingestion of a high carbohydrate meal
Breathe hydrogen concentration | 3 weeks
  Measurement of hydrogen in exhaled air as an indicator of carbohydrate absorption

REFERENCES:
- [Result] Augustin LSA, Kendall CWC, Jenkins DJA, Willett WC, Astrup A, Barclay AW, Bjorck I, Brand-Miller JC, Brighenti F, Buyken AE, Ceriello A, La Vecchia C, Livesey G, Liu S, Riccardi G, Rizkalla SW, Sievenpiper JL, Trichopoulou A, Wolever TMS, Baer-Sinnott S, Poli A. Glycemic index, glycemic load and glycemic response: An International Scientific Consensus Summit from the International Carbohydrate Quality Consortium (ICQC). Nutr Metab Cardiovasc Dis. 2015 Sep;25(9):795-815. doi: 10.1016/j.numecd.2015.05.005. Epub 2015 May 16. PMID 26160327
- See also: WHO Global Report on Diabetes — https://apps.who.int/iris/bitstream/handle/10665/204871/9789241565257_eng.pdf;jsessionid=6CEFCE5876A8E46F48B90A0FAEFFBF9B?sequence=1